CLINICAL TRIAL: NCT03710681
Title: Safety, Tolerability and Pharmacokinetics Studies Following Multiple Subcutaneous Injections of SHR-1314 in Adults With Moderate-to-severe Plaque Psoriasis
Brief Title: A Safety Study of Multiple Subcutaneous (s.c.) Injections of SHR-1314 in Adults With Moderate-to-severe Plaque Psoriasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1314-103
Record Dates: First submitted 2018-09-06; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Moderate-to-severe Plaque Psoriasis
Keywords: SHR-1314 Phase 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Multiple subcutaneous injections of SHR-1314 at 160mg every two weeks
  Interventions: Biological: SHR-1314
- Cohort 2 (Experimental): Multiple subcutaneous injections of SHR-1314 at 240mg every two weeks
  Interventions: Biological: SHR-1314

INTERVENTIONS:
Biological: SHR-1314 — Pharmaceutical form: Injection solution. Route of administration: subcutaneous injection.

SUMMARY:
This is a multiple dose escalating and open labeled clinical trial to evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple subcutaneous (s.c.) injections of SHR-1314 in adults with moderate-to-severe plaque psoriasis.

The primary objective of this study is to investigate the safety and tolerability of multiple doses of subcutaneous SHR-1314 in subjects with moderate-to-severe plaque psoriasis. Secondary objectives are to determine the pharmacokinetics (PK) and immunogenicity profile of SHR-1314 in subjects with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
16 subjects with 2 dose groups will be enrolled in the study, all of whom received the SHR-1314 without placebo control. There are 8 subjects in each cohort. The dose will be started at 160mg and will be escalated by following dose escalating rules. The primary endpoint is the safety and tolerability : adverse events, vital signs, physical examination, laboratory examination, 12 lead electrocardiogram, injection site reactions, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at age between 18 and 65 years old at screening.
2. History of chronic plaque-type psoriasis for at least 6 months, with either documented medical history of psoriasis for at least 6 months or confirmation of the diagnosis by the Investigator at screening, if the subject was diagnosed by another physician.
3. At the time of randomization, moderate to severe plaque psoriasis, defined by:

   * PASI score of 12 or greater and
   * PGA score of 3 or greater and
   * BSA affected by plaque-type psoriasis of 10% or greater.
4. A subject is a candidate for systemic psoriasis therapy and/or phototherapy and/or chemo phototherapy.
5. Body Mass Index (BMI) of 18 to 35 kg/m2 (inclusive) at screening.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic, and guttate psoriasis) at screening.
2. Drug-induced psoriasis (i.e. new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) at randomization.
3. Active systemic infections (other than common cold) during the two weeks before randomization (e.g., hepatitis), or serious infections requiring hospitalization and/or intravenous injection of antibiotic treatment within eight weeks prior to randomization.
4. History of inflammatory bowel disease or have other ongoing active autoimmune diseases.
5. At screening, history or symptoms of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
6. History of depression and/or suicidal ideation or any suicidal behavior based on clinical assessment by the investigator.
7. Have a known allergy or hypersensitivity to any biologic therapy at screening that would pose an unacceptable risk to the subject if participating in this study.
8. Are currently enrolled in, or discontinued from a clinical trial involving an IP within the last 4 weeks or at least 5 half-lives of the last dosing prior to randomization, whichever is longer; or concurrently enrolled (at randomization) in any other trials.
9. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test at screening or Day 0.
10. Females of childbearing potential (defined as all females physiologically capable of becoming pregnant) and males who are unwilling or unable to use highly effective contraception during the study and 21 weeks after the last administration of IP (anticipated 5 half-lives).
11. History of alcohol or illicit drug abuse within the year prior to screening.
12. Have any other condition that precludes the subject from following and completing the protocol, in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-04-21 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events [Safety and tolerability] | Baseline to 168 days after first dose administration
  Incidence and severity of adverse events, change from baseline in vital signs and 12-lead electrocardiogram.
Incidence of development of Anti-drug Antibodies (ADAs) [Safety and Tolerability] | Baseline to 168 days after first dose administration
  Incidence of development of Anti-drug Antibodies (ADAs) during the course of the study.

SECONDARY OUTCOMES:
Assessment of PK parameter | Baseline to 168 days after first dose administration
  time to maximum concentration (tmax)
Assessment of PK parameter | Baseline to 168 days after first dose administration
  maximum concentration (Cmax)
Assessment of PK parameter | Baseline to 168 days after first dose administration
  area under curve (AUC0-14days)
Assessment of development of Anti-drug Antibodies (ADAs) | Baseline to 168 days after first dose administration
  Incidence of development of Anti-drug Antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huanshan Hospital , Shanghai Fudan University, Shanghai, Shanghai Municipality
  - Huanshan Hospital , Shanghai Fudan University, Shanghai